CLINICAL TRIAL: NCT02334566
Title: Lending a Hand to Our Future: Documenting, Assessing and Treating Posttraumatic Stress Disorder in Refugee Children and Youth
Brief Title: Lending a Hand to Our Future: PTSD in Refugee Children and Youth
Acronym: LHOF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to complete study according to protocol
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 06705
Record Dates: First submitted 2014-12-30; First posted 2015-01-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Refugee children mental health; community health care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NET TX (Experimental): Behavioral intervention for PTSD (NET/KIDNET) with 8-12 sessions administered on a weekly basis.
  Interventions: Behavioral: NET TX
- Delayed TX (Active Comparator): Behavioral intervention for PTSD (NET/KIDNET) with 8-12 sessions administered on a weekly basis, started following a three-month wait period
  Interventions: Behavioral: NET TX

INTERVENTIONS:
Behavioral: NET TX — Intervention procedures are a behavioral intervention (NET & KIDNET) with 8-12 sessions administered on a weekly basis.

SUMMARY:
Immigrant and refugee children and youth are the fastest growing segment of Canadian society, but their mental health is too often overlooked even though their high rates of symptoms are increasingly of concern. These children and youth face the same developmental challenges as other children, but migration and resettlement amplify challenges and also create additional risks. Although a literature about the effects of immigrant family life on the mental health of children exists, very little research has examined the specific extent and implications of post-traumatic stress disorder (PTSD) among refugee children and youth. In addition, the best practice intervention strategies that most optimally support their mental health difficulties have not been evaluated. This study investigates the effectiveness of a treatment intervention in a sample of refugee children: Narrative Exposure Therapy or NET and KIDNET (developed for younger children), selected due to their documented superiority relative to other forms of treatment for children and youth with PTSD.

DETAILED DESCRIPTION:
Refugee children and youth are at high risk for post-traumatic stress disorder (PTSD) and related psychological distress potentially interfering with optimal adjustment and development in the host country. Following extensive efforts and a workshop by the Partnership for Health System Improvement Initiative, comprised of researchers, decision makers, practitioners, immigrant service agencies and related community groups in Ontario, it was determined that research addressing this at-risk population is a priority area. The current study addresses this urgent need by aiming to enhance the health system's capacity in relation to the needs of one of Canada's most vulnerable population. As local refugee settlement continue to rise and reported rates for PTSD in refugee children and youth remain startling; often intensified by historical traumatic factors such as the intensity of exposure to war and other atrocities prior to migration, it is essential to research this highly vulnerable population. In particular, a need exists for research, such as the current study, that specifically documents, assesses and treats PTSD in refugee children and youth, thereby increasing knowledge in the community and preventing further negative outcomes by improving education and health care systems. Although treatment interventions exist for PTSD, the many unique challenges faced by refugee populations are often overlooked. Narrative Exposure Therapy (NET or KIDNET), designed to restore agency and provide symptom relief, is one intervention for PTSD treatment that can indicate positive outcomes for refugee populations. The current proposal describes a research study to address the needs of this at-risk population through pilot testing of the feasibility of providing PTSD intervention within two school-based primary health care programs and an inner city youth shelter in Toronto. The results will contribute to our understanding of the feasibility of a model of intervention, which can be made available for use in other jurisdictions of Ontario and across Canada to improve adjustment and prevent mental health problems.

This is research project will utilize a randomized clinical trial of treatment for PTSD. It includes refugee children and youth, between the ages of 7 and 15, from two established MHSPI clinics, which currently serve approximately 40 schools, with a total school-aged population of more than 20,000 as well as youth between the ages of 16 and 19 from Covenant House. This study will draw on established measures for PTSD mental health and trauma histories through the use of standardized rating scales and interview methods. Interpreters will be made available and sensitivity adjustments for language and culture will be made. Research assistants will be trained to administer the UCLA screening instruments for PTSD to identify potential contributing or mediating factors of outcome . In addition, paediatricians will be trained in the UCLA diagnostic process to provide case identification, and graduate/medical students will be trained in NET/KIDNET, to facilitate implementation and evaluation of the treatment procedures. All children and youth enrolled at the two MSPHI and Covenant House clinics will placed into one of 3 groups: 'refugee', 'other immigrant' and 'native-born', and be screened for PTSD. All study participants, with a score of 15 or higher, as recommended by the UCLA group, will then be included in the next phase which consists of in depth clinical assessment. Of these participants who are identified as PTSD diagnostic cases are then included in the treatment evaluation phase: randomized into the control- treatment groups and placed into gender-paired therapeutic dyads, i.e. female therapists will be paired with female children and adolescents with PTSD and males with males. Ten male and 10 female therapists will take part in the project and each will be assigned to treat 20 people with PTSD, resulting in a total estimated treated study sample of 400. The control group participants will proceed to the exact same treatment procedures following a three-month wait. All participants included in the treatment groups, either immediate or waiting list control, will receive 3, 6 and 12 month follow-up assessments to evaluate PTSD symptoms using the same UCLA measurements to screen initially. All data will be collected, coded and analyzed using standard statistical analyses appropriate to the research design.

ELIGIBILITY:
Inclusion Criteria:

* All referrals, to the school-based health centers (SBHC) at Parkdale and Sprucecourt schools, through the school support team (SST), individual teachers, parents or community contacts.
* SBHC children and youth between the ages of 7 and 16 years of age
* All referrals to Covenant House for youth between 16 and 18 years of age (up to 19th birthday)
* Assessed to qualify for either Refugee status or Immigrant status, and who request participation and consent to research procedures
* Participants with a score of 15 or higher on UCLA PTSD-RI and are case identified (diagnosed) by paediatricians for PTSD

Exclusion Criteria:

* Participants with a score on the UCLA-PTSD-RI lower than 15.
* Participants with a score on the UCLA-PTSD-RI higher than 15 and diagnosed with PTSD by paediatrician
* Participants identified as native born
* Participants with known (previously identified) disorders that impact on communication and/or cognition, such as Developmental Disability, Autism, Communication Disability.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 588 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in UCLA-PTSD-RI (UCLA-Posttraumatic Stress Disorder-Reaction Index) | week 1, week 12, week 24, week 48, week 64
  Although treatment interventions exist for PTSD, the many unique challenges faced by refugee populations are often overlooked. Narrative Exposure Therapy (NET or KIDNET), designed to restore agency and provide symptom relief, is one intervention for PTSD treatment that can indicate positive outcomes for refugee populations.

CONTACTS AND LOCATIONS:
Overall Officials: Morton Beiser, M.D., Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No
Dataset is incomplete and not usable